CLINICAL TRIAL: NCT04880837
Title: Human Papillomavirus Education Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Electra Paskett, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OSU-20370; NCI-2021-00730 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-05-06; First posted 2021-05-11 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Human Papillomavirus-Related Carcinoma
MeSH Terms: interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prevention (educational session, handout, survey) (Experimental): Participants attend educational session about HPV-related cancers, screening, and HPV vaccination and guidelines and receive informational infographic handout on HPV vaccination. Participants also complete surveys pre and post education session over 5 minutes each to assess HPV vaccination status among children of participants, HPV knowledge, and intentions to get the HPV vaccination, and screening among participants. In addition, participants complete surveys over telephone or face-to-face at 3 and 6 months.
  Interventions: Other: Educational Intervention; Other: Informational Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Educational Intervention — Attend educational session
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Informational Intervention — Receive handouts
Other: Survey Administration — Complete surveys

SUMMARY:
This clinical trial aims to implement a culturally-tailored educational outreach actives with the goal of increasing knowledge of human papillomavirus (HPV) types that can lead to cancer and uptake of the available vaccine. The initiative also addresses barriers to vaccination and refer people to sites where they can get the HPV vaccine (e.g., private doctor offices, community health clinics, school-based health centers, and health departments). The HPV education program may help increase HPV vaccination rates and ultimately prevent HPV-related cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To implement culturally tailored educational outreach activities with the goal of increasing knowledge of HPV types that can lead to cancer and uptake of the available vaccine.

OUTLINE:

Participants attend educational session about HPV-related cancers, screening, and HPV vaccination and guidelines and receive informational infographic handout on HPV vaccination. Participants also complete surveys pre and post education session over 5 minutes each to assess HPV vaccination status among children of participants, HPV knowledge, and intentions to get the HPV vaccination, and screening among participants. Participants participate in surveys over telephone or face-to-face at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* From Ohio

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in human papillomavirus (HPV) knowledge | Baseline up to 6 months
  Change in knowledge and strength of intention to be vaccinated will be correlated with key outcomes, specifically actual vaccination and actions promoting vaccination (e.g., encouraging HPV vaccination with family/friends, talking to their doctor/provider about the HPV vaccine). Multivariable logistic regression analyses will be conducted to examine the impact of knowledge change and strength of intentions on these binary outcomes (vaccinated/not vaccinated and encouraged/did not encourage HPV vaccination) controlling for important covariates such as age, sex, race/ethnicity, education, primary language, and health insurance/health care coverage.

CONTACTS AND LOCATIONS:
Overall Officials: Electra D Paskett, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu